CLINICAL TRIAL: NCT05875259
Title: A Randomized, Open-label, Multiple-dose, 6-sequence, 3-treatment, 3-period, Crossover Study to Evaluate the Pharmacokinetic Interaction and Safety Between BR1019-1 and BR1019-2 in Healthy Adult Subjects
Brief Title: A Clinical Trial Study to Evaluate the Pharmacokinetic Interaction and Safety Between BR1019-1 and BR1019-2 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FDC-CT-101
Record Dates: First submitted 2023-05-11; First posted 2023-05-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 1: A-B-C
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2
- Sequence 2 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 2: A-C-B
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2
- Sequence 3 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 3: B-A-C
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2
- Sequence 4 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 4: B-C-A
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2
- Sequence 5 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 5: C-A-B
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2
- Sequence 6 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 6: C-B-A
  Interventions: Drug: BR1019-1; Drug: BR1019-2; Drug: BR1019-1 + BR1019-2

INTERVENTIONS:
Drug: BR1019-1 — Treatment group A : One tablet of BR1019-1 administered alone once daily for 7 days.
Drug: BR1019-2 — Treatment group B : One tablet of BR1019-2 administered alone once daily for 7 days.
Drug: BR1019-1 + BR1019-2 — Treatment group C : One tablet each of BR1019-1 and BR1019-2 administered in combination once daily for 7 days.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interaction and safety between BR1019-1 and BR1019-2 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 55 years at screening
* Those who voluntarily decide to participate in the study and provide written consent to follow the study directions after listening to and fully understanding the detailed explanation on this study

Exclusion Criteria:

* Those who have clinically significant diseases associated with the cardiovascular system, respiratory system, liver, kidney, nervous system, endocrine system, blood/tumor, psychiatric disorders, or urinary system, as well as drug abuse, or a history thereof.
* Those who took any prescription drugs or herbal medicines within 14 days prior to the first day of administration or any over-the-counter (OTC) drugs within 7 days prior to the first day of administration (however, if other conditions are appropriate according to the judgment of the investigator, they may participate in the clinical study.)
* Those who took drugs inducing and inhibiting drug-metabolizing enzymes, such as barbiturates, within 30 days prior to the study initiation.
* Those who have been on a diet (especially grapefruit juice or its products) that may affect the absorption, distribution, metabolism, and excretion of the drug within 7 days prior to the first day of administration.
* Pregnant women, potentially pregnant women, or breast-feeding women Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using medically acceptable methods of contraception* throughout the entire period from the date of the first administration of the investigational product to the end of the clinical study

  * Medically acceptable methods of contraception: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used
* Those who are unwilling or unable to comply with the dietary and lifestyle guidelines required for the clinical study
* Those who have clinically significant abnormalities in the results of other clinical laboratory tests or who have been determined by the investigator to be ineligible to participate in the clinical study due to other reasons (e.g., non-compliance with instructions, uncooperative attitude, etc.)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
AUC0-24,ss | 0-48 hours after administration
  Area under the concentration-time curve from 0 h to 24 h of BR1019-1 and BR1019-2 at steady-state
Cmax,ss | 0-48 hours after administration
  Maximum concentration of drug in plasma of BR1019-1 and BR1019-2 at steady-state

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No